CLINICAL TRIAL: NCT04066868
Title: Evaluating the Use of Patient-Reported Outcome Measures for Improving the Inter-Rater Reliability of Common Terminology Criteria for Adverse Event Ratings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Collaborators: Bezirkskrankenhaus Kufstein (Unknown); Centre Hospitalier Universitaire de Besancon (Other); Martin-Luther-Universität Halle-Wittenberg (Other); Università di Cagliari (Unknown); Kansai Medical University (Other); King Hussein Cancer Center (Other); Tata Memorial Hospital (Other Government); Rigshospitalet, Denmark (Other); Clinical Hospital Center Rijeka (Other); N.N. Blokhin National Medical Research Center of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1020/2019
Record Dates: First submitted 2019-08-19; First posted 2019-08-26 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Cancer
Keywords: patient-reported outcomes (PRO); common terminology criteria for adverse events (CTCAE); quality of life; electronic data assessment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRO active (Experimental)
  Interventions: Other: Patient-reported outcomes assessment; Other: CTCAE rating; Other: PRO data is displayed
- PRO not active (Active Comparator)
  Interventions: Other: Patient-reported outcomes assessment; Other: CTCAE rating

INTERVENTIONS:
Other: Patient-reported outcomes assessment — Patient-reported outcomes are electronically assessed using EORTC QOL measures
Other: CTCAE rating — CTCAE Ratings are conducted by clinicians
Other: PRO data is displayed — PRO data is displayed right next to the CTCAE rating
  Arms: PRO active

SUMMARY:
This open randomized trial investigates, if clinicians complete CTCAE ratings differently when receiving patients' patient-reported outcome (PRO) data prior to their CTCAE completion. The primary objective is to demonstrate superior inter-rater reliability of CTCAE ratings from physicians relying on EORTC PRO data as additional data source over traditional CTCAE ratings not including PRO information.

DETAILED DESCRIPTION:
In oncology, detection and tracking of adverse events (AEs) are a top priority in both clinical trials and routine care. The classification of AEs mostly relies on the Common Toxicity Terminology for Adverse Events (CTCAE) developed by the US-American National Institutes of Health and the National Cancer Institute.

It is known, however, that the assessment of AEs can greatly vary depending on whether they are assessed by patients or by clinicians.

Procedure: The patients (any oncological diagnosis, day clinic or inpatient for treatment with chemotherapy or immunotherapy; open 1:1 randomized) fill out an EORTC quality of life questionnaire electronically (C30 + further questions). These PRO data are immediately available for the clinicians. Independently of each other, two different clinicians conduct a medical consultation with the patient and electronically a CTCAE rating. For the intervention Group, clinicians see the PRO values directly next to the input options for the CTCAE rating. For the control Group, clinicians see the input options for the CTCAE rating. The similarity of the assessments is checked using intra-class correlation.

The combined use of PROs and CTCAE data makes particular sense for AEs/aspects that are directly experienced by the patient (fatigue, pain, cognitive problems, emotional functioning, ...) and can only be adequately recorded by the clinician through communication with the patient.

ELIGIBILITY:
Inclusion Criteria:

* any Cancer diagnosis
* current treatment with chemotherapy or immunotherapy
* symptom burden equal or greater score 3 of the screening question "On a scale of 0 to 10, to what degree did you experience physical or emotional symptoms/problems during the last week?"
* ability to understand the questions linguistically and cognitively
* written informed consent

Exclusion Criterion:

* psychiatric diagnosis or mental health problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1013 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
EORTC Quality of Life Questionnaire C30 and additional questions from the EORTC Item Library | single assessment of quality of life before the medical consultation
  patient-reported quality of life
CTCAE V5.0 | single assessment during the medical consultation with physician 1 on the same day of PRO assessment
  physician 1 rates patient symptoms (17 CTCAE domains matching the EORTC C30 and additional questions)
CTCAE V5.0 | single assessment during the medical consultation with physician 2 on the same day of PRO assessment
  physician 2 rates patient symptoms (17 CTCAE domains matching the EORTC C30 and additional questions)

CONTACTS AND LOCATIONS:
Locations (1):
- Bezirkskrankenhaus Kufstein, Kufstein, Austria

REFERENCES:
- [Derived] Wintner LM, Sztankay M, Abdel-Razeq H, Hamdan-Mansour R, Caocci G, Mouillet G, Kikawa Y, Shibata N, Krishnamurthy MN, Joshi A, Krishnatry R, Jain A, Pappot H, Petranovic D, Trobentar A, Schmidt H, Schulze S, Tararykova A, Zabernigg A, Giesinger JM, Holzner B; EORTC Quality of Life Group. Inter-rater reliability of CTCAE assessments with or without EORTC patient-reported outcome data in a mixed cancer population: a multinational, open-label, randomised controlled trial. Lancet Oncol. 2026 Jan 19:S1470-2045(25)00679-5. doi: 10.1016/S1470-2045(25)00679-5. Online ahead of print. PMID 41570841
- [Derived] Wintner LM, Giesinger JM, Sztankay M, Bottomley A, Holzner B; EORTC Quality of Life Group. Evaluating the use of the EORTC patient-reported outcome measures for improving inter-rater reliability of CTCAE ratings in a mixed population of cancer patients: study protocol for a randomized controlled trial. Trials. 2020 Oct 13;21(1):849. doi: 10.1186/s13063-020-04745-w. PMID 33050917
- See also: Study protocol publication — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-020-04745-w